CLINICAL TRIAL: NCT04074460
Title: Volatile Anaesthesia and Perioperative Outcomes Related to Cancer (VAPOR-C): A Feasibility Study
Brief Title: Volatile Anaesthesia and Perioperative Outcomes Related to Cancer Feasibility Study
Acronym: VAPOR-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Melbourne Health (Other); The Alfred (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 16/144
Record Dates: First submitted 2019-08-15; First posted 2019-08-30 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Cancer, Breast; Cancer Colorectal; Cancer Prostate; Cancer, Lung; Cancer Melanoma Skin; Cancer, Other
Keywords: major surgeries lasting >2 hours
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Melanoma; Neoplasms | interventions — Propofol; Isoflurane; Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients are blinded to the anaesthetic type given. Statistician also blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (TIVA) (Active Comparator): Propofol-based total intravenous anaesthesia
  Interventions: Drug: Propofol
- Volatile (Active Comparator): Volatile-based (isoflurane, sevoflurane or desflurane) general anaesthesia
  Interventions: Drug: isoflurane, sevoflurane or desflurane

INTERVENTIONS:
Drug: Propofol — General Anaesthesia
  Arms: Propofol (TIVA)
Drug: isoflurane, sevoflurane or desflurane — General Anaesthesia
  Arms: Volatile

SUMMARY:
A multicentre, prospective randomized, active-controlled feasibility trial of volatile-based anaesthesia vs. propofol-based total intravenous anaesthesia to investigate the impact of anaesthesia on long-term (i.e. 5-years) patient cancer outcomes in patients undergoing elective major cancer surgery.

DETAILED DESCRIPTION:
This study aims to assess the feasibility of conducting a phase IV, multi-centre, single-blinded, randomized control trial (VAPOR-C (Main)).

Primary aims To measure the ability to recruit eligible patients into the study.

To measure the ability to successfully deliver each of the two anaesthetic techniques (volatile-based general anaesthesia and propofol-based anaesthesia) according to the research protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-80 years
* Elective surgery
* Major cancer surgery expecting to last two or more hours, for:
* Breast (mastectomy or segmentectomy plus sentinel node dissection)
* Colorectal
* Lung
* Prostate
* Melanoma (excision of melanoma plus lymph node dissection AND/OR skin flap construction
* Other major cancer surgeries (e.g. oesophagectomy, head and neck cancer, etc.)

Exclusion Criteria

* Palliative surgery for end-stage disease with no curative intent
* Emergency surgery
* Extensive comorbid disease, i.e. American Society of Anesthesiologists (ASA) Score > 4
* Age <18 or >80 years old
* Refusal or inability to provide valid informed consent
* Risk of severe postoperative nausea and vomiting (PONV risk score >3)
* Previous allergy or contraindication to either anaesthetic medication
* Indication for gas induction of anaesthesia
* Currently enrolled in another clinical trial unless agreed by the coordinating principal investigator and site principal investigator that co-enrolment can occur.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2017-08-27 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
To measure the ability to recruit eligible patients into the study. | 18 months
  The study protocol will be assessed as feasible if a recruitment rate of at least 75% is achieved.
To measure the ability to successfully deliver each of the two anaesthetic techniques (volatile-based general anaesthesia and propofol-based anaesthesia) according to the research protocol. | 18 months
  The study protocol will be assessed as feasible if a successful delivery rate of at least 90% is achieved.

SECONDARY OUTCOMES:
To identify that all sites can capture data within the electronic case report form (eCRF) and utilize the electronic data capturing system (REDCap). | 18 months
  All missing data to be recorded including reason for missing data, where available. Quantitative and qualitative analysis of reasons for missing data will be analysed by : Number of fields with missing data (percentage) and reason for missing data ( qualitative descriptor). Fields with >1 missing data point will be analysed for reasons for failure.
To test the efficiency of the centralized patient enrolment and computer randomization system. | 18 months
  Number of events of failed randomisation will be recorded on eCRF (under 'treatment of subjects"). Quantitative analysis of failed randomisation (reported as %) as well as descriptive reason for failure will be recorded and analysed. This will allow shortcomings in the use of the computer-generated centralised randomisation program to be identified and ratified.

CONTACTS AND LOCATIONS:
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No